CLINICAL TRIAL: NCT02363413
Title: Initiation of Non- Invasive Ventilation at Home Versus Hospital Among Patients With Overlap Syndrome: Randomized Controlled Non-inferiority Study
Brief Title: Initiation of Non- Invasive Ventilation at Home Versus Hospital Among Patients With Overlap Syndrome
Acronym: OVNI-Dom
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IP Santé Domicile (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VNI_001
Record Dates: First submitted 2015-01-27; First posted 2015-02-16 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Overlap Syndrome
Keywords: NIV; Overlap Syndrom; home; hospital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IniVAH (Active Comparator): Initiation of the NIV in hospital : current care. 3 days hospitalization to start-up the NIV as usual.
  Interventions: Other: IniVAH
- IniVAD (Experimental): Initiation of the NIV at home : experimental care.
  Interventions: Other: IniVAD

INTERVENTIONS:
Other: IniVAH — Initiation of the NIV during a 3 days hospitalization as usual.
  Other Names: Initiation of the NIV at hospital : current care
  Arms: IniVAH
Other: IniVAD — Initiation of the NIV at home. The first day, the kinesiologist and the technician start-up the NIV at home with the patient. The investigator will validate the adjustment settings proposed by the kinesiologist. No procedure during the second day as described by the HAS. The third day, the kinesiologist and the technician come back to the patient home so as to adjust the settings if needed and if validated by the investigator.
  Other Names: Initiation of the NIV at home
  Arms: IniVAD

SUMMARY:
The study is based on the assumption that in the Overlap Syndrome, the introduction at home of the NIV is as effective in terms of compliance and clinical and gazometric improvement, and life quality, that setting hospital start up. The investigators will study the initiation of NIV at home versus in hospital in two randomized Overlap Syndrome patient groups. The main objective of the study is to demonstrate the non-inferiority of the initiation of the NIV at home versus hospital in terms of compliance.

DETAILED DESCRIPTION:
The Overlap Syndrome is defined by the coexistence of chronic obstructive pulmonary disease (COPD) and an apnea - hypopnea syndrome obstructive sleep (SAHS). The interaction between these two diseases is responsible for deepest nocturnal desaturation, decreased sensitivity to CO2, more pronounced sleep alterations, more frequent daytime hypercapnia, a higher risk of hypertension pulmonary and increased cardiovascular risk, compared to subjects with COPD or isolated SAHS.

The Overlap Syndrome treatments are continuous positive airway pressure (CPAP) or non-invasive ventilation (NIV), associated complemented or not by oxygen therapy during sleep. The criteria for choosing the type of treatment are not well defined. Quality and compliance of the NIV are very important in all diseases leading to chronic respiratory failure whose Overlap Syndrome. The increase in the number of patients treated with NIV is estimated at over 12% per year. The NIV startup is usually performed in a conventional hospitalization but congestion healthcare pathways lead to increase waiting time before treatment. Thus, to date, no study has validated a supported alternative to meet the increase in the number of patients on NIV while maintaining quality service.

The HAS has defined good candidates for a NIV home based startup, on the following criteria: patients with a recognized indication of NIV in the long term , with stable respiratory failure, requiring only nocturnal ventilation, surrounded by caregivers mastering the use of equipment and whose location allows rapid intervention. The study is based on the assumption that in the Overlap Syndrome, the introduction at home of the NIV is as effective in terms of compliance and clinical and gazometric improvement, and life quality, that setting hospital start up. The investigators will study the initiation of NIV at home versus in hospital in two randomized Overlap Syndrome patient groups. The main objective of the study is to demonstrate the non-inferiority of the initiation of the NIV at home versus hospital in terms of compliance.

ELIGIBILITY:
Inclusion Criteria:

* Major patients, of less than 80 years
* Patients with chronic respiratory failure within a Overlap syndrome ( defined by the coexistence of COPD and OAS ) in stable situation (no exacerbation for at least 4 weeks) , indication for a NIV treatment
* OAS confirmed by polysomnography according to the standards of the American Academy of Sleep Medicine ( AASM ) with an AHI> 15, the central apneas are tolerated if < 20%
* COPD defined by obstruction of the air flow : VEMS/CVF <70 % and VEMS <80% of the average value predicted
* Started criteria of NIV: chronic respiratory failure within an Overlap Syndrome and PaCO2 > 45 mmHg (at rest on room air ) and / or medium PtCO2 > 50 mmHg
* Patient informed of the study and who signed an informed consent

Exclusion Criteria:

* Patients already treated for OAS in the year
* Patient tracheotomised
* Other diseases with respiratory involvement : neuromuscular disease , restrictive disease of the chest with CPT <80% , apnea syndrome pure central sleep ( central apnea are tolerated if < 20% )
* Lung cancer within the last 5 years
* Uncontrolled psychic diseases
* Acute respiratory failure requiring NIV , going back a month
* Clinical situation requiring prolonged hospitalization
* Patients with no opportunity to understand and follow instructions
* Refusal to participate in the study
* Lack of insurance coverage
* Pregnant and / or nursing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
compliance- average adherence measured over the three months under NIV expressed in hours/night | month 3 (M3)

SECONDARY OUTCOMES:
quality of ventilation : evolution of the pCO2 and nocturnal saturation at M3 | month 3 (M3)
quality of life and satisfaction of the patients : patient life satisfaction questionnaire | month 3 (M3)
the occurrence of complications : number of NIV complication occurred | month 3
economic study- number of hospitalization nights | month 3 (M3)
economic study- number of intervention of the kinesiologist and the technician | month 3 (M3)
economic study- number of phone contact by the patient | month 3 (M3)

CONTACTS AND LOCATIONS:
Overall Officials: Safia Maaradji-Gati, MD, Study Director — IPSanté Domicile; Jésus Gonzalez, MD, Principal Investigator — La Pitié-Salpétrière; Marie Pia D'orthor, MD, Principal Investigator — Hôpital Bichat - Claude Bernard
Locations (17):
- France (17):
  - CH Annecy-Genevois, Annecy
  - Clinique Chirurgicale Bel-Air, Bordeaux
  - CH Cannes, Cannes
  - CHU Dijon, Dijon
  - CH Intercommunal du Val d'Ariège, Foix
  - Hôpital Raymond Poincaré, Garches
  - CHU de Grenoble site Nord - Hôpital Albert Michallon, Grenoble
  - Centre Hospitalier Haguenau, Haguenau
  - Clinique Du Blanc Mesnil, Le Blanc-Mesnil
  - Clinique Mutualiste du Medoc, Lesparre-Médoc
  - CHR - Hôpital Calmette, Lille
  - CHU Bichat - Claude Bernard, Paris
  - CHU La Pitié-salpétrière, Paris
  - Clinique Saint Laurent, Rennes
  - Institut Arnault Tzanck, Saint-Laurent-du-Var
  - CHU de Strasbourg - Hôpital Civil, Strasbourg
  - Hôpital Larrey CHU Toulouse, Toulouse